CLINICAL TRIAL: NCT05333536
Title: Effects of Strength Training on Freestyle Swimming Performance and Core Muscles Strength in Swimmers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0424 Nayab
Record Dates: First submitted 2022-02-20; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Sports Physical Therapy
Keywords: Stroke rate; Free style; Stability ball; Core strength

STUDY DESIGN:
Intervention Model Description: Two groups , comparison group a control and b experimental
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group exercises (Experimental): Experimental performs Strengthening exercises of core.10 reps , 3 sets of each.Prone plank(10 sec hold)(18) ,Side plank (8 sec hold),Bridging (8 sec hold)(19),Bird dog (10 reps ,3 sets),Leg drop (10 reps, 3 sets)(15),Dying bug with their regular swimming practice. First 2 weeks simple strengthening exercises.Next 4 weeks stability ball exercises. Dying bug without stability ball. And strengthening exercises of UL and LL with theraband ,10 reps each.Upper limb: Latissimus dorsi,Serratus anterior, Upper trapezius.Lower Limb: Flexors of hip, Extensors of hip,Plantar flexors.
  Interventions: Other: Experimental: Experimental group exercises
- Control group (Active Comparator): control only participates in their yearly swimming trainings.
  Interventions: Other: No Intervention: Control group

INTERVENTIONS:
Other: Experimental: Experimental group exercises — Experimental performs Strengthening exercises of core.10 reps , 3 sets of each.Prone plank(10 sec hold)(18) ,Side plank (8 sec hold),Bridging (8 sec hold)(19),Bird dog (10 reps ,3 sets),Leg drop (10 reps, 3 sets)(15),Dying bug with their regular swimming practice. First 2 weeks simple strengthening exercises.Next 4 weeks stability ball exercises. Dying bug without stability ball. And strengthening exercises of Upper Limb and Lower Limb with theraband ,10 reps each.Upper Limb: Latissimus dorsi,Serratus anterior, Upper trapezius.Lower limb : Flexors of hip, Extensors of hip,Plantar flexors.
  Arms: Experimental group exercises
Other: No Intervention: Control group — control only participates in their yearly swimming trainings.
  Arms: Control group

SUMMARY:
To compare the effectiveness performance and core muscles of Strength Training . strength in swimmers on freestyle swimming

DETAILED DESCRIPTION:
There is lack of literature on strength training on freestyle swimming performance, core muscles strength in swimmers, kicking, and stroke rate. With the help of this study the swimming performance of individual s will improve.

ELIGIBILITY:
Inclusion Criteria:

* Competitive swimmers
* male gender
* Experience of more than a year of swimming

Exclusion Criteria:

* Individuals with associated neuromuscular conditions and any injuries to lower limbs.
* Spinal injuries have been excluded in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male swimmers will participate
Enrollment: 18 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
50 meter Swimming Test | 6th week
  Done by stop watch, changes will be assessed accordingly: First week Pre test and post test in 6th week which will be last week of work
Core muscle strength test | 6th week
  Determine by stop watch .Used for monitoring of core strength of athlete. There are 8 levels Level 1: plank position hold for 60sec, Level 2: right arm lift and hold for 15 sec, Level 3: left arm lift for 15 sec, Level 4: right leg lift for 15 sec, Level 5: left leg lift for 15 sec, Level 6: right arm and left leg lift from floor for 15 secs, Level 7: left arm and right leg lift from floor for 15 sec, Level 8: then again hold plank for 30 sec. If individual feel difficulty at some level then end the test, and record that level. Good = complete, Poor= unable to perform.
  Changes will be assessed accordingly: First week Pre test and post test in 6th week which will be last week of work
Stroke rate | 6th week
  Firstly calculate time need to complete three 3 stroke cycles. Then evaluate stroke rate by using this formula. SR= 60 × 3/tSR (SR- Stroke Rate, tSR- time taken of 3 cycles) Changes will be assessed accordingly: First week Pre test and post test in 6th week which will be last week of work
Kicking | 6th Week
  Time need for 50 meter of kicking performance by the use of kickboard ,stop watch use.
  Changes will be assessed accordingly: First week Pre test and post test in 6th week which will be last week of work
Manual muscle testing (mmt) grading scale 0-5 | 6th Week
  Latissimus dorsi, Serratus anterior,Upper trapezius,Flexors of hip,Extensors of hip,Plantar flexors by grading 0=no contraction,1= flickering contraction,2=full range of motion eliminated gravity,3= full range of motion against gravity,4= full range of motion with minimal resistance,5= full range of motion against maximal resistance Changes will be assessed accordingly: First week Pre test and post test in 6th week which will be last week of work

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, Principal Investigator — Riphah International University
Locations (1):
- Punjab international swimming complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eskiyecek CG, Gül M, Uludağ B, Gül GK. The Effect of 8-Week Core Exercises Applied to 10-12 Age Male Swimmers on Swimming Performance. International Journal of Applied Exercise
- [Background] Gencer YG. Effects of 8-Week Core Exercises on Free Style Swimming Performance of Female Swimmers Aged 9-12. Asian Journal of Education and Training. 2018;4(3):182-5.
- [Background] Marani IN, Subarkah A, Hermawan I, Pradana VO. Core Exercise To Strengthen The Core Muscle for Swimming.
- [Background] Heinlein SA, Cosgarea AJ. Biomechanical Considerations in the Competitive Swimmer's Shoulder. Sports Health. 2010 Nov;2(6):519-25. doi: 10.1177/1941738110377611. PMID 23015983
- [Background] Moser C, Sousa CV, Olher RR, Nikolaidis PT, Knechtle B. Pacing in World-Class Age Group Swimmers in 100 and 200 m Freestyle, Backstroke, Breaststroke, and Butterfly. Int J Environ Res Public Health. 2020 May 30;17(11):3875. doi: 10.3390/ijerph17113875. PMID 32486151
- [Background] Sawdon-Bea J, Benson J. The effects of a 6-week dry land exercise program for high school swimmers. Journal of physical education and sports management. 2015;2(1):1-17.
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Fig G. Strength training for swimmers: Training the core. Strength & Conditioning Journal. 2005;27(2):40-2.
- [Background] Venâncio BO, Tacani PM, Deliberato PCP. Pain prevalence in swimming athletes of São Caetano do Sul. Revista Brasileira de Medicina do Esporte. 2012;18:394-9.
- [Background] Gatta G, Cortesi M, Di Michele R. Power production of the lower limbs in flutter-kick swimming. Sports Biomech. 2012 Nov;11(4):480-91. doi: 10.1080/14763141.2012.670663. PMID 23259238
- [Background] Schneider P, Meyer F. Anthropometric and muscle strength evaluation in prepubescent and pubescent swimmer boys and girls. Revista Brasileira de Medicina do Esporte. 2005;11:209-13
- [Background] Morouco PG, Marinho DA, Amaro NM, Pérez-Turpin JA, Marques MC. Effects of dry-land strength training on swimming performance: a brief review. Journal of Human Sport and Exercise. 2012;7(2):553-9
- [Background] Gönener A, Gönener U, Yılmaz O, Horoz T, Demirci D. The effect of 8-week thera-band exercises on male swimmers' 100 m freestyle swimming performance. Journal of Human Sciences. 2017;14(4):3950-5
- [Background] Patil D, Salian SC, Yardi S. The effect of core strengthening on performance of young competitive swimmers. International Journal of Science and Research. 2014;3(6):2470-7.
- [Background] Weston M, Hibbs AE, Thompson KG, Spears IR. Isolated core training improves sprint performance in national-level junior swimmers. Int J Sports Physiol Perform. 2015 Mar;10(2):204-10. doi: 10.1123/ijspp.2013-0488. Epub 2014 Jul 8. PMID 25025936
- [Background] Mujik a I, Crowley E. Strength training for swimmers. Concurrent Aerobic and Strength Training: Springer; 2019. p. 36986.
- [Background] Amara S, Barbosa TM, Negra Y, Hammami R, Khalifa R, Chortane SG. The Effect of Concurrent Resistance Training on Upper Body Strength, Sprint Swimming Performance and Kinematics in Competitive Adolescent Swimmers. A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Sep 29;18(19):10261. doi: 10.3390/ijerph181910261. PMID 34639560
- [Background] Atkins SJ, Bentley I, Brooks D, Burrows MP, Hurst HT, Sinclair JK. Electromyographic response of global abdominal stabilizers in response to stable- and unstable-base isometric exercise. J Strength Cond Res. 2015 Jun;29(6):1609-15. doi: 10.1519/JSC.0000000000000795. PMID 26010796
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] Patel RS, Sharma A, Prajapati U, Dave V, Varma M. Effect of Strength Training on Performance of Young Competitive swimmersA Randomized Control Trial.
- [Background] Avers D, Brown M . Daniels and Worthingham's Muscle Testing, First South Asia Edition E Book: Techniques of Manual Examinationand Performance Testing: Elsevier; 2018.